CLINICAL TRIAL: NCT00872924
Title: An Open Label, Bioequivalence Study of Sumatriptan Succinate 100 mg Tablets (Containing 140 mg of Sumatriptan Succinate Equivalent to 100 mg Sumatriptan) Under Fasting Conditions
Brief Title: Bioequivalence Study of Sumatriptan 100mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 219_SUMAT_08
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sumatriptan succinate 100 mg tablets (containing 140 mg of sumatriptan succinate equivalent to 100 mg sumatriptan) of OHM laboratories Inc. (A subsidiary of Ranbaxy Pharmaceuticals Inc., USA).
  Interventions: Drug: sumatriptan 100mg
- 2 (Active Comparator): IMITREX® 100 mg tablets (containing 140 mg of sumatriptan succinate equivalent to 100 mg sumatriptan)
  Interventions: Drug: sumatriptan 100mg

INTERVENTIONS:
Drug: sumatriptan 100mg

SUMMARY:
An open label, bioequivalence study of sumatriptan succinate 100 mg tablets (containing 140 mg of sumatriptan succinate equivalent to 100 mg sumatriptan) under fasting Conditions

DETAILED DESCRIPTION:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioequivalence study comparing Sumatriptan Succinate Tablets 100 mg (containing sumatriptan succinate equivalent to 100 mg sumatriptan) manufactured by OHM Laboratories Inc. with IMITREX® tablets 100 mg (containing sumatriptan succinate equivalent to 100 mg sumatriptan) manufactured by GlaxoSmithkline Research Triangle Park, NC 27709, Made in Canada in healthy, adult, male, human subjects under fasting condition.

Following an overnight fast of at least 10 hour, a single oral dose of sumatriptan succinate tablets 100 mg (containing 140 mg of sumatriptan succinate equivalent to 100 mg sumatriptan) of either test or reference formulation was administered during each period of the study, along with 240 mL of drinking water at ambient temperature under low light condition and supervision of trained study personnel.

32 subjects were enrolled into the study. However, twenty seven (27) subjects completed both the periods of the study. Pharmacokinetic and Statistical analysis was performed on twenty seven subjects (27) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Were in the age range of 18-45 years.
2. Were neither overweight nor underweight for their height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Had voluntarily given written informed consent to participate in this study.
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

1. Had history of known hypersensitivity to Sumatriptan or related group of drugs or to any other drug.
2. Had history of intermittent chest pain and or chest tightness which might or might not require medication for relief.
3. Had history of peripheral vascular disease (cramping, tiredness and or severe pain on walking relatively shorter distances persisting on rest, noticeable change in color (blueness or paleness) or temperature (coolness) when compared to the other limb).
4. Had history of headache, vertigo, dizziness with or without nausea vomiting.
5. Had history of intermittent loss of vision.
6. Had history of seizure and or head injury.
7. Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
8. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
9. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for hemoglobin, total white blood cells count, differential WBC count or platelet count.
10. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
11. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
12. Had clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
13. Had clinically abnormal ECG or Chest X-ray.
14. Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma head-injury or coma.
15. Had history of any psychiatric illness which might impair the ability to provide written informed consent.
16. Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
17. Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
18. Used of any enzyme modifying drugs within 30 days prior to Day 1 of the study.
19. Participation in any clinical trial within 12 weeks preceding Day 1 of the study.
20. Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Ranbaxy Sumatriptan 100mg tablets under fasting conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy CPU, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html